CLINICAL TRIAL: NCT05804916
Title: A Single-center, Blinded, Efficacious, Phase III Randomized Clinical Trial Initiated by Investigators to Investigate the Use of Surface Guided Radiation Therapy (SGRT) in Combination With Deep Inspiration Breath Hold (DIBH) Technique for Left Breast Cancer Treatment, Compared to Traditional Laser Alignment With Free Breathing Treatment
Brief Title: Optical Surface Monitoring Technology-Guided Large-Segment Radiotherapy for Breast Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGRT-BC
Record Dates: First submitted 2023-03-13; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer; Optical Surface Monitoring Technology; Large-segment Radiotherapy
Keywords: breast cancer; optical surface monitoring technology; large-segment radiotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Control group: Patients with left breast cancer treated with traditional laser alignment with a free breathing treatment Study group: Patients with left breast cancer treated with SGRT combined with the DIBH technique
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SGRT+DIBH group (Experimental): Patients with left breast cancer treated with SGRT combined with DIBH technique
  Interventions: Device: Surface Guided Radiation Therapy (SGRT)
- common+Free breath group (No Intervention): Patients with left breast cancer treated with traditional laser alignment with free breathing treatment

INTERVENTIONS:
Device: Surface Guided Radiation Therapy (SGRT) — SGRT and DIBH those two devices could be combined together to improve the accuracy in radiation therapy position and heart protection
  Other Names: Deep Inspiration Breath Hold (DIBH) technique
  Arms: SGRT+DIBH group

SUMMARY:
This study is a single-center,blinded, efficacious, phase III randomized clinical trial initiated by investigators. The primary objective is to investigate the use of Surface Guided Radiation Therapy (SGRT) in combination with Deep Inspiration Breath Hold (DIBH) technique for left breast cancer treatment, compared to traditional laser alignment with free breathing treatment. This approach offers superior positioning accuracy and improved heart protection without any increase in radiation or adverse reactions.

DETAILED DESCRIPTION:
This is an investigator-initiated blinded, efficacious, phase III randomized clinical trial study. The study hypothesis is that the use of Surface Guided Radiation Therapy (SGRT) in combination with the Deep Inspiration Breath Hold (DIBH) technique for left breast cancer treatment can improve positioning accuracy and heart protection without any increase in radiation or adverse reactions. The primary endpoint of this study is the accuracy of the treatment location and incidence of patient coronary events/myocardial perfusion decline.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have undergone breast-conserving surgery or modified radical mastectomy for left breast cancer;
2. Planned whole-breast ± supraclavicular region, chest wall ± supraclavicular region radiotherapy;
3. Able to perform deep inspiration breath-hold technique with breath-holding time >35s and can repeat it continuously for more than 6 times;
4. Patients who have not received neoadjuvant chemotherapy or breast reconstruction surgery;
5. No active heart disease, myocardial infarction, congestive heart failure or other cardiac diseases at baseline;
6. Patients are fully voluntary and able to sign the informed consent form 30 days before enrollment.

Exclusion Criteria:

1. Bilateral breast cancer;
2. No pathological diagnosis;
3. Remote metastasis;
4. Receiving neoadjuvant chemotherapy or breast reconstruction;
5. Have received mediastinal radiotherapy in the past;
6. Previous history of abdominal or pelvic radiotherapy;
7. Previous or secondary primary malignant tumor;
8. Serious cardiac insufficiency; Myocardial infarction or uncorrected unstable arrhythmia or uncorrected unstable angina pectoris occurred in the last 3 months; Pericardial disease.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — aged 18-70, with an expected lifespan of >5 years
Enrollment: 556 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of treatment location | Change from baseline to the whole treatment procedure
  surface optical monitoring technology and simulation of surface contour registration error generated by surface optical surface error, as well as errors obtained by Cone beam CT registration. The translational errors in the left-right (x), up-down (y), front-back (z) directions, and rotational errors Rx, Ry, Rz will be measured
Incidence of patient coronary events/myocardial perfusion decline | 3-year
  including the cardiac enzymes, ECG and myocardial perfusion

SECONDARY OUTCOMES:
Secondary efficacy indicators | 3-year
  Correlation between surface optical monitoring technology and CBCT offset values Correlation between positioning errors and dose pass rates Patient position movement within fractions
cardiac safety | 5-year
  cardiac injury events include myocardial enzymes, electrocardiogram, echo, etc
patients' quality of life | 5-year
  scale scores of EORTC-QLQ-BR23, 0-100 scores, higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided